CLINICAL TRIAL: NCT06220552
Title: Low-dose Radiotherapy Combined With Sintilimab and Temozolomide in Recurrent Glioblastoma: A Single-arm, Prospective Phase II Clinical Study
Brief Title: The Efficacy and Safety of Low-dose Radiotherapy Combined With Sintilimab and Temozolomide in Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yingpeng Peng, Director, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.TJBZLK.003
Record Dates: First submitted 2024-01-13; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — sintilimab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-dose Radiotherapy Combined With Sintilimab and Temozolomide (Experimental)
  Interventions: Drug: Sintilimab; Radiation: Low-dose Radiotherapy

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg D1, Q3W
Radiation: Low-dose Radiotherapy — Radiotherapy 1Gy/1F, D1/D2/D8/D15, Q3W

SUMMARY:
This is an open-label, single-arm, phase II clinical trial to explore the efficacy and safety of low-dose radiotherapy combined with programmed death 1 (PD-1) inhibitor (sintilimab) and temozolomide in recurrent glioblastoma. The eligible patients are scheduled to administered sintilimab 200mg D1 Q3W temozolomide 50mg/m2 QD and radiotherapy 1Gy/1F D1/D2/D8/D15 Q3W for 4-6 cycles, then sintilimab for maintenance. The overall primary study hypothesis is that the combination regimen of low-dose radiotherapy, sintilimab and temozolomide is safe and feasible in the treatment of recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed glioblastoma, radiographically or pathologically diagnosed recurrence.
2. Aged ≥ 18 years.
3. ≥12 weeks after postoperative radiotherapy.
4. Karnofsky performance status (KPS) ≥ 60.
5. Expected survival > 3 months.
6. Adequate organ function, based on meeting all of the following criteria (no blood components and cytologic growth factors were received within 14 days prior to the test):

   1. Hemoglobin ≥ 90 g/L; absolute neutrophil count ≥ 1.5 × 10^9/L; and platelet count ≥ 100 × 10^9/L;
   2. Serum albumin ≥ 28 g/L;
   3. Total bilirubin ≤ 1.5 × upper limit of normal (ULN); Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN;
   4. Serum creatinine ≤ 1.5 × ULN;
   5. Activated partial clotting enzyme time and international standardized ratio (INR) ≤ 1.5 × ULN (Patients on stable doses of anticoagulant therapy such as low molecular weight heparin or warfarin with INR within the expected treatment range of anticoagulants can be screened ).
   6. Thyroid stimulating hormone ≤ ULN; If abnormal, T3 and T4 levels should be examined, and if T3 and T4 levels are normal, they can be screened.
7. Subjects voluntarily join the study and sign an informed consent form, with good compliance.

Exclusion Criteria:

1. Treatment with a dose of prednisone > 10mg /d or equivalent dose of corticosteroids is required.
2. There exist other uncontrolled central nervous system diseases unrelated to cancer.
3. A history of other malignant tumors within the previous 5 years or at the time of enrollment, except for cured skin basal cell carcinoma and cervical in situ cancer, as well as thyroid papilloma.
4. Uncontrolled cardiac clinical symptoms or diseases, such as New York Heart Association (NYHA) class II or above heart failure, unstable angina pectoris, myocardial infarction within 1 year, patients with clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention.
5. Serious infections, such as severe pneumonia, bacteremia, and infection comorbidities requiring hospitalization, occurred within 4 weeks.
6. Active autoimmune diseases, such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; It does not include patients with vitiligo or childhood asthma/allergies that have healed and require no intervention as adults.
7. A history of immunodeficiency, including HIV-positive status or other acquired congenital immunodeficiency diseases, or a history of organ transplantation and bone marrow transplantation.
8. Patients with active tuberculosis infection found by history or CT examination, or patients with active tuberculosis infection history within 1 year prior to enrollment, or patients with active tuberculosis infection history before 1 year without formal treatment.
9. Active hepatitis B (HBV DNA ≥ 2,000 IU/mL or 10,000 copies/mL) or hepatitis C (positive HCV antibody test and HCV RNA above the lower limit of detection).
10. Known history of psychotropic drug abuse, alcoholism and drug use.
11. Not suitable for inclusion, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | from the first day of treatment to the follow up of 1 year
  median progression free survival

SECONDARY OUTCOMES:
overall survival (OS) | from the first day of treatment to the follow up of 1 year
  median overall survival
Adverse events | from the first day of treatment to the follow up of 1 year
  CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Yingpeng Peng, Zhuhai, Guangdong, China